CLINICAL TRIAL: NCT06926140
Title: Effectiveness of Acupuncture Combined With PD-1/PD-L1 Inhibitors for Advanced Lung Cancer：A Randomized Controlled Clinical Study
Brief Title: Acupuncture Combined With PD-1/PD-L1 Inhibitors for Advanced Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Liu Zhishun, professer，Chief Physician, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-195-KY
Record Dates: First submitted 2025-03-31; First posted 2025-04-13 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-05

CONDITIONS: Lung Cancers
Keywords: lung cancer; acupuncture; immunotherapy
MeSH Terms: conditions — Lung Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acupuncture (Experimental)
  Interventions: Device: Acupuncture
- sham acupuncture (Sham Comparator)
  Interventions: Device: Sham Comparator

INTERVENTIONS:
Device: Acupuncture — Both groups have a standard anti-tumor Western medical treatment regimen (PD-1/PD-L1 inhibitor combined with chemotherapy); the acupuncture group is combined with acupuncture treatment. The day of starting antitumor treatment for each cycle was D1; D1-D5 was performed by the investigator on the patient for 2 times of acupuncture treatment, once a day; D8-D13 and D15-D20 were operated by patients or family members, and the investigator remotely assisted via video to complete the press needle treatment 4 times each, once a day, for four consecutive synergistic cycles, for a total of 24 times. The main acupuncture points are Guanyuan (Ren Mai 4), Shangyintang (EX-HN3), Taiyang (EX-HN5), Taichong (Liv-3), Zusanli (ST-36), and Xin (CO-15).
  Arms: Acupuncture
Device: Sham Comparator — Both groups have a standard anti-tumor Western medical treatment regimen (PD-1/PD-L1 inhibitor combined with chemotherapy); the sham acupuncture group is combined with sham acupuncture treatment. The day of starting antitumor treatment for each cycle was D1; D1-D5 was performed by the investigator on the patient for 2 times of sham acupuncture treatment, once a day; D8-D13 and D15-D20 were operated by patients or family members, and the investigator remotely assisted via video to complete the sham press needle treatment 4 times each, once a day, for four consecutive synergistic cycles, for a total of 24 times. The main acupuncture points are Guanyuan (Ren Mai 4), Shangyintang (EX-HN3), Taiyang (EX-HN5), Taichong (Liv-3), Zusanli (ST-36), and Xin (CO-15).
  Other Names: sham acupuncture
  Arms: sham acupuncture

SUMMARY:
This study will be an evaluation of the efficacy and safety of acupuncture to enhance the response rate of immunotherapy in advanced lung cancer. The main questions it aims to answer are 1. Does acupuncture heighten the response rate of immunotherapy in advanced lung cancer? 2. Does acupuncture heighten the safety of immunotherapy in advanced lung cancer? Researchers will compare acupuncture to sham acupuncture to see if acupuncture could enhance the response rate of immunotherapy in advanced lung cancer. Both groups will receive a standard anti-tumor Western medical treatment regimen (PD-1/PD-L1 inhibitor combined with chemotherapy), and the experimental and control groups will be treated with 4 cycles of acupuncture or sham-acupuncture on top of the anti-tumor treatment regimen, respectively. Patients were followed up every three weeks for the first three months and every three months thereafter to record any disease progression, adverse events, survival or mortality status, and so on.

ELIGIBILITY:
Inclusion criteria:

* Age 18-75 years;
* ECOG/PS score of grade 0-1 and expected survival ≥ 3 months;
* Non-small cell lung cancer AJCC lung cancer staging of stage IIIB-IV, or small cell lung cancer staging of extensive stage;
* PD-L1 immunohistochemistry detection of tumor cell positive proportion score (TPS) <50%;
* Non-small cell lung cancer adenocarcinoma patients do not have EGFR-sensitive mutations, ALK fusions, ROS1 fusions, BRAFV600 mutations, NTRK fusions, RET fusions, MET14 skipping mutations, and amplified gene-driven mutations by genetic testing;
* Patients with no previous systemic therapy/first-line treatment;
* Patients suitable for chemotherapy combined with immunotherapy;
* Traditional Chinese Medicine (TCM) diagnosis of Qi Depression;
* Having at least 1 measurable tumor lesion (diameter > 1cm) or lymph node short diameter ≥ 1.5cm;
* Sign the informed consent form and voluntarily participate in this study.

Exclusion criteria:

* Combined with other primary malignant tumors;
* Those who have contraindications to immunotherapy after basic assessment of immunotherapy;
* Those with autoimmune diseases or those who need long-term treatment with systemic steroids or immunosuppressants;
* Those with combined serious and uncontrolled primary diseases of heart, cerebrovascular, liver, kidney, hematopoietic system and so on;
* Those with metal allergy or severe fear of needles;
* Those who are pregnant or breastfeeding;
* Those who are unable to cooperate to complete the assessment due to mental disorder, intellectual or language impairment;
* Those with active severe infectious or inflammatory diseases;
* Those who have received acupuncture treatment or other clinical trials within 1 month prior to randomization;
* In the judgment of the investigator, persons who have a concomitant medical condition that seriously jeopardizes the safety of the participant or interferes with the completion of the study, or who are deemed to have other reasons for not being suitable for enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-06-21 (Actual); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | At 0,4,7,10,13 weeks,6,9,12,15,18,21,24 months from randomization, until progression occurred

SECONDARY OUTCOMES:
Disease Control Rate | At 0,4,7,10,13 weeks,6,9,12,15,18,21,24 months from randomization, until progression occurred
Progression-Free Survival | At 0,4,7,10,13 weeks,6,9,12,15,18,21,24 months from randomization, until progression occurred
Overall Survival | At 0,4,7,10,13 weeks,6,9,12,15,18,21,24 months from randomization, until death occurred.
Eastern Cooperative Oncology Group Performance Status, ECOG PS | At 0,4,7,10,13 weeks,6,9,12,15,18,21,24 months from randomization, until death occurred
  Levels 0 to 5, the lower the level, the better the physical condition.
GAD-7 | At 0,4,7,10,13 weeks,6 months from randomization
  The total score range is 0-21 points, higher scores indicates worse results.
PHQ-9 | At 0,4,7,10,13 weeks,6 months from randomization
  The total score range is 0-27 points, higher scores indicates worse results.
Insomnia Severity Index | At 0, 4, 7, 10, and 13 weeks and 6 and 9 months from randomization
  The total score range is 0-28 points, higher scores indicates worse results.
Lung Cancer Symptom Scale | At 0,4,7,10,13 weeks,6,9 months from randomization
  Each item is scored using the Visual Analog Scale (0-100mm), with higher scores indicating more severe symptom burden.
weight | At 0,4,7,10,13 weeks,6,9,12,15,18,21,24 months from randomization, until progression or death occurred
adverse event | At 0,4,7,10,13 weeks,6,9,12,15,18,21,24 months from randomization, until progression or death occurred
  Collect blood routine, liver function, kidney function, thyroid function, myocardial enzyme spectrum, incidence of adverse reactions, and immune therapy related adverse reactions. Record the type, grading, correlation with treatment, start and end time of adverse reactions
Duration of immunotherapy | At 0,4,7,10,13 weeks,6,9,12,15,18,21,24 months from randomization, until immunotherapy is no longer used

OTHER OUTCOMES:
Assessment of belief in acupuncture | Baseline assessment (week 0)
  Participants will be asked: Do you think your lung cancer may be helped by acupuncture?
Blinding assessment | Within 5 minutes after either treatment at week 10.
  Participants will be asked: Do you think you have received traditional acupuncture in the past 10 weeks?

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Guang'anmen Hospital, Chinese Academy of Traditional Chinese Medicine, Beijing, Beijing Municipality
  - Hunan Provincial Integrated Traditional Chinese and Western Medicine Hospital, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data and data dictionary will be available with the publication until six months after publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Deidentified participant data and data dictionary will be available with the publication until six months after publication.
Access Criteria: A formal request should be sent to zhishunjournal@163.com with a methodologically sound proposal.